CLINICAL TRIAL: NCT03364907
Title: Clinical pharmacoloGy of platinUm-based hyperThermic Intraperitoneal Chemotherapy: Exploration of the Impact of Flushing on tumOur, Systemic and Personnel eXposure (GUTOX)
Brief Title: Clinical Pharmacology of Platinum-based Hyperthermic Intraperitoneal Chemotherapy
Acronym: GUTOX
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: GUTOX
Record Dates: First submitted 2017-10-02; First posted 2017-12-07 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-07

CONDITIONS: Peritoneal Carcinomatosis
Keywords: HIPEC; oxaliplatin; flushing; peritoneal carcinomatosis
MeSH Terms: conditions — Peritoneal Neoplasms; Flushing | interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — peritoneal tissue samples, blood samples, instillate samples and wound exudate samples will be collected from the patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HIPEC patients: Patients with a diagnosis of peritoneal carcinomatosis who undergo HIPEC treatment with oxaliplatin.
  Interventions: Other: HIPEC with flushing afterwards; Other: HIPEC without flushing afterwards

INTERVENTIONS:
Other: HIPEC with flushing afterwards — flushing with saline fluid after HIPEC
Other: HIPEC without flushing afterwards — NO flushing with saline fluid after HIPEC

SUMMARY:
Currently, there is a lack of knowledge on the effect of additional flushing after HIPEC on tumour platinum exposure, systemic platinum exposure and platinum concentration in drain exudate and thereby personal exposure. Therefore the investigators want to perform a study to investigate the effect of flushing after HIPEC on tumour exposure, systemic exposure and on wound exudate concentration.

DETAILED DESCRIPTION:
Cytoreductive surgery combined with hyperthermic intraperitoneal chemotherapy (HIPEC) is standard care in the treatment of patients with peritoneal carcinomatosis as a result of intra-abdominal cancers. In many (inter)national centres oxaliplatin is used for the primary HIPEC treatment. Although the oxaliplatin dose of 460mg/m2 is widely accepted, the exact procedure of HIPEC differs between institutions and surgeons. Due to a great variety in the volume of the abdominal cavity, platinum concentration in the perfusate might differ between patients. Moreover, there is no consensus about the usefulness of flushing the HIPEC system with crystalloids at the end of oxaliplatin administration. Flushing is predominantly performed with the idea to minimize both systemic exposure of ultrafilterable platinum and personnel exposure to platinum contaminated exudate. On the other hand, HIPEC without flushing might increase effectiveness because intraperitoneal tumour cells are exposed to high concentrations of oxaliplatin for a longer time period. The option of flushing is based on an individual preference of the surgeon. Currently, there is a lack of knowledge on the effect of flushing on tumour platinum exposure, systemic platinum exposure and platinum concentration in drain exudate and thereby personal exposure. Therefore the investigators want to perform a study to investigate the effect of flushing after HIPEC on tumour exposure, systemic exposure and on wound exudate concentration.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must provide written informed consent prior to performance of study-specific procedures or assessments and must be willing to comply with treatment and follow-up.

   Note: Informed consent may be obtained prior to start of the specified screening window.

   Note: Procedures conducted as part of the subject's routine clinical management (e.g., blood count, imaging study) and obtained prior to signing of informed consent may be utilized for screening or baseline purposes.
2. Age ≥ 18 years
3. Confirmed diagnosis of preoperatively identifi ed primary or recurrent peritoneal carcinomatosis (PC) of colorectal origin who are planned for HIPEC treatment with oxaliplatin according to routine clinical care

Exclusion Criteria:

1) Patients who do not achieve a cytoreduction score of CC-0 will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with peritoneal carcinomatosis who undergo HIPEC treatment with oxaliplatin as part of routine care.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-06-08 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
change in tissue platinum exposure before and after flushing | immediately after the oxaliplatin instillate solution is withdrawn from the abdominal cavity and immediately after additional flushing is performed. This takes all place within 1 hour after the start of HIPEC.
  Change in tissue platinum exposure of non-tumour peritoneal tissue sample before and after flushing with saline

SECONDARY OUTCOMES:
wound exudate platinum concentration | until day 3 post-HIPEC
  platinum concentration in wound exudate samples will be measured in the drains
systemic exposure of total and unbound platinum | until day 3 post-HIPEC
  systemic exposure of total and unbound platinum will be measured using 13 blood samples
total and unbound platinum concentration in instillate | all samples will be taken within 30 minutes during the HIPEC procedure
  total and unbound platinum concentration in instillate will be measured in 3 samples of instillate solution that will be obtained during the HIPEC procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] de Jong LAW, Elekonawo FMK, Lambert M, de Gooyer JM, Verheul HMW, Burger DM, de Wilt JHW, Chatelut E, Ter Heine R, de Reuver PR, Bremers AJA, van Erp NP. Wide variation in tissue, systemic, and drain fluid exposure after oxaliplatin-based HIPEC: results of the GUTOX study. Cancer Chemother Pharmacol. 2020 Jul;86(1):141-150. doi: 10.1007/s00280-020-04107-y. Epub 2020 Jun 27. PMID 32594200
- See also: paper — https://pubmed.ncbi.nlm.nih.gov/32594200/

DOCUMENTS (1):
  • Study Protocol (2017-11-16): https://cdn.clinicaltrials.gov/large-docs/07/NCT03364907/Prot_000.pdf